CLINICAL TRIAL: NCT04918212
Title: Safety and Efficacy Study of Fabulous Stent Graft System for Stanford B Aortic Dissection: A Prospective, Multi-center, Single Arm, Objective Performance Criteria Clinical Trial
Brief Title: Safety and Efficacy Study of Fabulous Stent Graft System for Stanford B Aortic Dissection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Endonom Medtech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WQ1601
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Aortic Dissection Type B

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fabulous Stent Graft System (Experimental): All patients received endovascular surgery using fabulous stent graft system
  Interventions: Device: Fabulous Stent Graft System

INTERVENTIONS:
Device: Fabulous Stent Graft System — All patients received endovascular surgery using fabulous stent graft system

SUMMARY:
A prospective, multi-center, objective performance criteria clinical trial to evaluate the safety and efficacy of Fabulous Stent Graft System manufactured by Hangzhou Endonom Medtech Co., Ltd. for Stanford B Aortic Dissection.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years old;
2. The informed consent was signed by the patient or the legal representative;
3. Diagnosed with Stanford B aortic dissection;
4. The proximal anchoring area of is 18-42 mm in diameter, and not less than 15mm in length;
5. Has a suitable arterial approach and is suitable for surgical treatment.

Exclusion Criteria:

1. The patient's distal vascular false cavity has been completely thrombotic or organized;
2. Pregnant or breastfeeding ;
3. Has participated in clinical trials of other devices ；
4. History of aortic surgery or endovascular repair surgery ;
5. Allergic to contrast agents and anesthetics ;
6. Allergic to stents or conveyors ;
7. Patients with true or false aortic aneurysm;
8. History of myocardial infarction, TIA or cerebral infarction within the past 3 months;
9. Life expectancy is less than 12 months;
10. Other situations in which the investigator judges that not suitable for endovascular treatment .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2017-11-25 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2020-10-13 (Actual)

PRIMARY OUTCOMES:
Number of patients with no incidence of major surgical or device related adverse events rate | within 30 days after surgery
  Surgical or device related major adverse events (MAE) : death, respiratory failure, renal failure, stroke, paraplegia, intestinal ischemia, cardiovascular and vascular complications caused by surgery or device
Clinical success rate | 12 months after surgery
  Clinical success is defined as : no displacement of Stent Graft System, no type I or III endoleak requiring treatment, no enlargement of the false lumen, thrombosis of the false lumen, and no rupture of the dissection

SECONDARY OUTCOMES:
adverse event rate | within 12 months after surgery
Immediate delivery success rate | immediately after the surgery
  The stent graft system was successfully transported to the correct position and released successfully
Immediate operation successful rate | immediately after the surgery
  After the operation, angiographic observation showed that the proximal covered stent was in an appropriate position and adhered well without obvious endoleak, while the distal bare stent was in an appropriate position and adhered well
Endoleak rate | within 12 months after surgery
Secondary surgical treatment rate | within 12 months after surgery
  Secondary endovascular or surgical treatment due to stent displacement, endoleak, or related complications after stent implantation

CONTACTS AND LOCATIONS:
Locations (24):
- China (24):
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Chinese People's Liberation Army General Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Xiangya Hospital of Central South University, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Hainan Provincial People's Hospital, Haikou
  - Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Anhui Provincial Hospital, Hefei
  - The First Affiliated Hospital of Kunming Medical College, Kunming
  - Liuzhou Workers' Hospital, Liuchow
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Jiangsu Provincial People's Hospital, Nanjing
  - The First Affiliated Hospital of Guangxi Medical University, Nanning
  - The Ninth People's Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai
  - The First Hospital of Hebei Medical University, Shijia Zhuang
  - Tianjin Medical University General Hospital, Tianjin
  - The First Affiliated Hospital of the Fourth Military Medical University, Xi'an
  - Yantai Yuhuangding Hospital, Yantai
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Henan Provincial People's Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No